CLINICAL TRIAL: NCT04500405
Title: Long-term Outcomes of Patients With Diverticulitis and Risk Factors for Recurrence: a Multi-center Cohort Study
Brief Title: Outcomes of Patients With Diverticulitis and Risk Factors for Recurrence
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202003113RINB
Record Dates: First submitted 2020-08-02; First posted 2020-08-05 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-01

CONDITIONS: Recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
In the Emergency Department (ED), patients with acute diverticulitis usually present with acute abdominal pain. Sometimes, or mostly, it is an exclusive diagnosis, meaning that the diagnosis would be made after other emergent and acute abdomens are excluded. The recurrent diverticulitis cost medical burden. The studies focusing on potential risk factors of recurrent diverticulitis, especially for those after an episode of acute diverticulitis, are limited.

DETAILED DESCRIPTION:
Diverticular disease of the colon is common in industrial countries and has significant impact on patient health as well as health care cost. It is common in both Western countries and some Asian countries. For example, in the past, colonic diverticulosis was rare in Japan; with detection rates as low as approximately 2% in 1960. The detection rate increased to approximately 20% in the 1980s and 1990s. Studies have reported that increasing rates of diverticulosis are caused by westernization of the diet in Asian countries and are becoming a medical concern. Diverticular disease-associated hospital admissions have risen steeply in the recent past, which are not completely accounted for by the increasingly aging population of western countries. Approximately 130,000 hospitalizations occurring every year in the United States are attributable to diverticular disease. An analysis of the age-adjusted hospitalization rate of diverticulitis in the United States showed an increase from 62 per 100,000 in 1998 to 76 per 100,000 in 2005. These admission rates increased most in younger patients (< 45 years old) and have remained unchanged in patients older than 65 years. In spite of low mortality rate in patients with acute diverticulitis, moderate to severe comorbidities occur in specific patient group.

Painter and Burkitt hypothesized it in their article in 1960s and 1970s. They based their hypothesis on the observation that individuals in different geographic locations such as western industrialized countries versus those in developing countries were noted to have different rates of prevalence. They postulated that those in industrialized nations tended to eat processed food that was low in fiber compared with individuals in Africa and Asia, where the disease was previously unknown.

The USA Health Professional study showed a higher risk of diverticulitis in men with higher body mass index (BMI), waist-to-hip ratio and waist circumference [8]. Obesity also significantly increases costs associated with management of the disease and its complications [9]. The effect of obesity on the risk of recurrent diverticulitis is unknown.

In the Emergency Department (ED), patients with acute diverticulitis usually present with acute abdominal pain. Sometimes, or mostly, it is an exclusive diagnosis, meaning that the diagnosis would be made after other emergent and acute abdomens are excluded. The recurrent diverticulitis cost medical burden. The studies focusing on potential risk factors of recurrent diverticulitis, especially for those after an episode of acute diverticulitis, are limited.

This is a retrospective cohort study conduct from Oct 2008 to Sep 2018. The patients were recruited from National Taiwan University Hospital (NTUH), NTUH Hsin-Chu Branch (HCH), and NTUH Yun-Lin Branch.

ELIGIBILITY:
Inclusion Criteria:

* the patients who (a) visited ED from Oct 2008 to Sep 2018; (b) were diagnosed as diverticulitis by computed tomography (CT); (c) were aged over 20.

Exclusion Criteria:

* the patients who (a) received CT at other hospital and lost image; (b) lost the follow-up after index ED admission.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who (a) visited ED from Oct 2008 to Sep 2018; (b) were diagnosed as diverticulitis by computed tomography (CT); (c) were aged over 20.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-05-31 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
recurrence after the first episode of diverticulitis | 5 years
  recurrence after the first episode of diverticulitis

SECONDARY OUTCOMES:
The diagnostic accuracy between the sonographic diagnosis and final diagnosis | one month
  The final diagnosis was referred to the diagnosis that two expert physicians reviewed the medical records

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Lien, Taipei, Taiwan